CLINICAL TRIAL: NCT07173998
Title: Prospective Observational Study on Quality of Life With Postoperative Atrial Fibrillation
Brief Title: Quality of Life in Patients With Postoperative Atrial Fibrillation After Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jakob Wollborn, MD, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2025P000238
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Atrial Fibrillation
Keywords: cardiac surgery; recovery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Target group: Adult patients undergoing cardiac surgery with cardiopulmonary bypass
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — SF-36, TSQM-9, qualitative questions

SUMMARY:
Prospective observational study on quality of life with postoperative atrial fibrillation after cardiac surgery using SF-36 and qualitative questions

DETAILED DESCRIPTION:
This is a prospective observational study on quality of life in patients after cardiac surgery with postoperative atrial fibrillation. Patients will answer surveys before their surgery as well as one and three months after their heart operation. The survey includes SF-36, TSQM-9 and qualitative questions.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* Ages 18-99 years old
* Scheduled to undergo cardiac surgery
* Able to answer survey questions

Exclusion Criteria:

* Persistent / permanent atrial fibrillation
* Atrial fibrillation at presentation for surgery
* Emergent operations

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 scores | before, one month and three months postop
  compare development and absolut SF-36 scores

SECONDARY OUTCOMES:
Qualitative questions | before, one month and three months postop
  exploratory evaluation of qualitative questions
TSQM-9 scores | one month and three months postop
  TSQM-9 scores in Afib-patients

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Wollborn, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No